CLINICAL TRIAL: NCT07280156
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study Assessing the Efficacy, Safety, and Dosing Regimen Selection of Multiple Intravenous Infusions of PRX-115 With and Without Methotrexate Versus Placebo in Adult Patients With Gout (RELEASE)
Brief Title: A Study to Investigate the Clinical Effect and the Safety of PRX-115 Infused Intravenously at Different Dosing Regimens, With and Without Methotrexate, Versus Placebo in Adults Gout Patients (RELEASE)
Acronym: RELEASE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB115-GT-201
Record Dates: First submitted 2025-12-03; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Gout
Keywords: gout; uricase; uric acid; hyperuricemia; PRX-115
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: Multiple IV infusions at a fixed dose per infusion, at different treatment intervals . For different dosing regimens, PRX-115 will be tested with and without the immunomodulator, MTX.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- E4W with placebo-MTX (Experimental): IV infusion of PRX-115 every 4 weeks (E4W) for a total of 6 doses with placebo-MTX
  Interventions: Biological: PRX-115; Other: Placebo-Methotrexate
- E4W with MTX (Experimental): IV infusion of PRX-115 every 4 weeks (E4W) for a total of 6 doses with MTX
  Interventions: Biological: PRX-115; Drug: Methotrexate (MTX)
- E6W with MTX (Experimental): IV infusion of PRX-115 every 6 weeks (E6W) for a total of 4 doses with MTX
  Interventions: Biological: PRX-115; Drug: Methotrexate (MTX)
- E8W with MTX (Experimental): IV infusion of PRX-115 every 8 weeks (E8W) for a total of 3 doses + 3 doses of PRX-115 placebo every alternating 8 weeks with MTX
  Interventions: Biological: PRX-115; Drug: Methotrexate (MTX)
- placebo E4W (Placebo Comparator): infusion of PRX-115 placebo every 4 weeks (E4W) for a total of 6 doses with placebo-MTX
  Interventions: Other: PRX-115 placebo; Other: Placebo-Methotrexate
- placebo E6W (Placebo Comparator): IV infusion of PRX-115 placebo every 6 weeks (E6W) for a total of 4 doses with placebo-MTX
  Interventions: Other: PRX-115 placebo; Other: Placebo-Methotrexate

INTERVENTIONS:
Biological: PRX-115 — intravenous (IV) infusion
  Arms: E4W with MTX; E4W with placebo-MTX; E6W with MTX; E8W with MTX
Drug: Methotrexate (MTX) — Oral MTX 15 mg weekly
  Arms: E4W with MTX; E6W with MTX; E8W with MTX
Other: PRX-115 placebo — intravenous (IV) infusion
  Arms: placebo E4W; placebo E6W
Other: Placebo-Methotrexate — Oral Placebo-MTX weekly
  Arms: E4W with placebo-MTX; placebo E4W; placebo E6W

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase II study assessing the efficacy, safety, and dosing regimen selection of multiple IV infusions of PRX-115 over 24 weeks, with or without MTX, versus the respective placebos in adult patients with gout.

DETAILED DESCRIPTION:
This study will evaluate the efficacy, safety, tolerability, immunogenicity, pharmacokinetics (PK), and pharmacodynamics (PD) of PRX-115 (a recombinant pegylated Uricase) in adult patients with gout. Participants will receive PRX-115 by intravenous (IV) infusions according to different treatment schedules, with and without the immunomodulator methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years of age.
2. Weight within the range of 50.0 - 150.0 kg.
3. Gout patients who failed to normalize sUA (<7 mg/dL) with or without xanthine oxidase inhibitors or uricosuric agent or have contraindications to these drugs.
4. Willing to discontinue any oral ULT
5. Females who are sterile, postmenopausal, or non-pregnant and using birth control methods.

Exclusion Criteria:

1. Any condition known to have arthritis as a clinical manifestation.
2. Positive testing for HBV,HCV, or HIV.
3. The patient is a pregnant or lactating female or plans to become pregnant during the study period.
4. Known allergy or sensitivity to the injected proteins, including pegylated products.
5. Prior exposure to any experimental or marketed uricase.
6. Patient treated with a medication known to have an influence on urate metabolism or clearance such as ULTs.
7. History of anaphylaxis, severe allergic reactions, or severe atopy.
8. G6PD deficiency or known catalase deficiency.
9. History of significant hematologic or autoimmune disorders within 5 years of Screening and/or patient is immunocompromised or treated with immunosuppressive medications.
10. Non-compensated CHF or hospitalization for CHF (Stage 3-4 NYHA Functional Class) within 3 months of the Screening Visit, uncontrolled arrhythmia, treatment for acute coronary syndrome (myocardial infarction or unstable angina), or uncontrolled BP (>160/100 mmHg) at screening and prior to randomization at Week -4 (Visit 1).
11. Current liver disease, as determined by ALT or AST levels above upper limit of normal at Screening Visit.
12. Chronic liver disease.
13. Hemoglobin <11 g/dL, neutrophil count <1500 /µl, or platelet count <100,000 /µl.
14. Known severe pulmonary fibrosis, bronchiectasis or interstitial pneumonitis.
15. eGFR ≤ 40 mL/min/1.73m2 tested at Screening Visit. Kidney transplant or requires dialysis.
16. Known intolerance and/or known contraindication to MTX treatment or MTX treatment considered inappropriate
17. Has uncontrolled type 2 diabetes at Screening with HbA1c ≥8.5%. Patients with type 1 diabetes will be excluded.
18. Has known latent autoimmune diabetes of adult.
19. Immunocompromised state, regardless of etiology.
20. History or treatment of malignancy in the last 5 years, excluding localized, nonmelanoma skin cancers (e.g. basal or squamous cell)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Serum Uric Acid (sUA) Responders (sUA < 6 mg/dL) During Month 6 | 6 months of treatment
  Proportion of patients who achieve a reduction in sUA to <6.0 mg/dL for at least 80% of the time during Month 6

SECONDARY OUTCOMES:
Percentage of Serum Uric Acid (sUA) Responders (sUA < 6 mg/dL) at different time points | 3 to 6 months of treatment
  Proportion of patients that achieve a reduction in sUA to <6.0 mg/dL for at least 80% of the time during Month 3 or 4, 5 and 6.
Safety of PRX-115 | From enrollment to 8 months of study
  Occurrence and severity of treatment-emergent adverse events (TEAEs)